CLINICAL TRIAL: NCT01438359
Title: A Single-centre, Open-label, Three-period Study of the Pharmacokinetic Effect of PA21 on Furosemide in Healthy Male and Female Adults
Brief Title: A Drug-Drug Interaction Study of Furosemide and PA21
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PA-DDI-002
Record Dates: First submitted 2011-09-16; First posted 2011-09-22 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Drug-drug interaction; Pharmacokinetics; PA21; Drug Interaction Potentiation
MeSH Terms: interventions — Furosemide; Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PA21 and Furosemide with food (Experimental)
  Interventions: Drug: PA21 and Furosemide with food
- No PA21; Furosemide with food (Experimental)
  Interventions: Drug: No PA21; Furosemide with food
- PA21 with food and Furosemide 2hrs later (Experimental)
  Interventions: Drug: PA21 with food and Furosemide 2hrs later

INTERVENTIONS:
Drug: PA21 and Furosemide with food — The maximum dose of PA21 will be 15.0 g/day. The maximum dose of Furosemide will be 40 mg/day
  Arms: PA21 and Furosemide with food
Drug: No PA21; Furosemide with food — The maximum dosage of Furosemide will be 40 mg/day
  Arms: No PA21; Furosemide with food
Drug: PA21 with food and Furosemide 2hrs later — The maximum dose of PA21 will be 15 g/day. The maximum dose of Furosemide will be 40 mg/day
  Arms: PA21 with food and Furosemide 2hrs later

SUMMARY:
The purpose of this study is to determine if Furosemide is affected by PA21.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written informed consent

Exclusion Criteria:

* No significant medical conditions
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Effect of PA21 on Furosemide | PK assessment on Day 0, 11, and 22: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48 hrs post furosemide dose
  To assess the effect, if any, of PA21 on Furosemide exposure(AUC0-24; AUC0-infinity; Cmax; Tmax and t1/2).

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Winkle, MD, Principal Investigator — ACRI - Phase 1 (Advanced Clinical Research Institute)
Locations (1):
- ACRI - Phase 1, Anaheim, California, United States